CLINICAL TRIAL: NCT03122899
Title: Study of Bone Growth in the Sacroiliac Joint After Minimally Invasive Surgery With Titanium Implants
Acronym: SALLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SI-BONE, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300243
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Sacroiliac Dysfunction
Keywords: SI-BONE; sacroiliac joint; degenerative sacroiliitis; sacroiliac joint disruption; iFuse

STUDY DESIGN:
Intervention Model Description: Minimally invasive sacroiliac joint fusion surgery with iFuse-3D
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SIJ fusion with iFuse 3D with 6 mo CT (Other): These subjects will get pelvic CT at 6 months post-operatively.
  Interventions: Device: SIJ fusion with iFuse-3D
- SIJ fusion with iFuse 3D with 12 mo CT (Other): These subjects will get pelvic CT at 12 months post-operatively.
  Interventions: Device: SIJ fusion with iFuse-3D

INTERVENTIONS:
Device: SIJ fusion with iFuse-3D — Minimally invasive SIJ fusion with iFuse-3D titanium implant (usually 3 implants per SIJ).

SUMMARY:
SALLY studies sacroiliac joint fusion with the iFuse-3D implant.

DETAILED DESCRIPTION:
Participants will all get sacroiliac joint fusion on this study using the iFuse-3D titanium implant, manufactured by SI-BONE, Inc. Participants will be followed for clinical outcomes at pre-planned time points on the trial. Participants will be randomized to CT scan at 6 months or 12 months, and all will also get a CT scan at 5 years, the final visit for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 21-70 at time of screening.
2. Patient has suspected SI joint pain for greater than or equal to 6 months inadequately responsive to conservative care.
3. Diagnosis of sacroiliac joint dysfunction on one or two sides to be treated on study that is a direct result of sacroiliac joint disruption and/or degenerative sacroiliitis and is based on ALL of the following:

   1. Patient has pain at or close to the posterior superior iliac spine (PSIS) with possible radiation into buttocks, posterior thigh or groin and can point with a single finger to the location of pain (Fortin Finger Test) (on any targeted side), and
   2. Patient has positive findings on at least 3 physical examination maneuvers that stress the target SI joint(s) and
   3. Patient has block on any study targeted side with improvement in SI joint pain numeric rating scale (NRS) at 30 or 60 minutes of at least 50% after injection of local anesthetic into any affected SI joint with an immediate pre-block NRS of at least 5.
4. Baseline Oswestry Disability Index (ODI) score of at least 30%.
5. Baseline (average over the last week) SI joint pain score of at least 50 on 0-100 mm visual analog scale on any side to be treated under the study.
6. Patient has signed study-specific informed consent form.
7. Patient has the necessary mental capacity to participate and is physically able to comply with study protocol requirements.
8. Patient's insurance coverage for SI joint treatment has been considered and plan is to submit all study-related healthcare to insurance (or it is the patient's responsibility) (any required preauthorization should be completed prior to randomization on study).
9. Investigator believes patient is appropriate candidate for surgery using iFuse-3D Implant.

Exclusion Criteria:

1. Patient has bilateral SI joint symptoms with VAS pain scores ³50 on both sides and patient refuses to undergo bilateral treatment according to the study protocol.
2. Patient is currently pregnant, actively trying to become pregnant or is planning to become pregnant in the next year.
3. Severe back or hip pain due to other causes, such as lumbar disc degeneration, lumbar disc herniation, lumbar spondylolisthesis, lumbar spinal stenosis, lumbar facet degeneration, lumbar vertebral body fracture, piriformis syndrome, femoral acetabular impingement, labral tear or hip osteoarthritis. Patients with low back pain VAS ratings more than 50 should be carefully considered; they should not participate if the investigator believes these non-SIJ conditions would impair improvement from SIJ treatment.
4. SI joint dysfunction due to an alternative explanation such as:

   1. Inflammatory sacroiliitis (e.g., ankylosing spondylitis or other HLA-associated spondyloarthropathy)
   2. Tumor
   3. Infection
   4. Acute or unstable fracture.
5. History of recent (<1 year) major non-pregnancy-related trauma to pelvis.
6. Surgeon believes patient body habitus prevents surgery.
7. Previously diagnosed osteoporosis (defined as prior T-score <-2.5 or history of osteoporotic fracture) or prior/current use of drug therapy for osteoporosis.
8. Prior fracture of any bone related to cancer/tumor (i.e., pathologic fracture).
9. Prior diagnosis of tumor in sacrum or ilium.
10. Unstable fracture of sacrum and or ilium involving the targeted SIJ.
11. Osteomalacia or other metabolic bone disease.
12. Diagnosed or suspected chronic rheumatologic condition (e.g., rheumatoid arthritis, lupus).
13. Any known condition or anatomical deformity or variation that makes treatment with the iFuse-3D Implant infeasible.
14. Any known health condition that could prevent long-term follow-up required in this study.
15. Known allergy to titanium or titanium alloys.
16. Use of medications known to have detrimental effects on bone quality and soft-tissue healing.
17. Current local or systemic infection that raises the risk of surgery.
18. Patient currently receiving or seeking short- or long-term worker's compensation related to the SI joint or low back pain, currently receiving disability remuneration related to SI joint or low back pain, and/or currently involved in injury litigation related to the SI joint or low back pain.
19. Patient is a prisoner or a ward of the state.
20. Patient has known or suspected active drug or alcohol abuse.
21. Patient is unwilling to sign the study-associated opioid contract.
22. Diagnosed uncontrolled psychiatric disease (e.g., schizophrenia, major depression, personality disorders) that could interfere with study participation.
23. Patient is participating in an investigational study or has been involved in an investigational study within 3 months prior to evaluation for participation.
24. Patient has known or suspected fibromyalgia.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Primary Radiographic Outcome: Bone adherence | Comparing 6 and 12 month CTs to historical data from other studies.
  Percent surface area of the sacral end of the implants to which bone is adherent.
Primary Clinical Outcome: Disability due to low back pain | Comparing baseline to 6 months.
  Improvement in Oswestry Disability Index

SECONDARY OUTCOMES:
Bridging Bone | 6 months, 12 months, and 5 years
  Proportion of treated SIJs with bridging bone.
Clinically Significant Radiolucency | 6 months, 12 months, and 5 years
  Proportion of treated SIJs with evidence of clinically significant radiolucency.
Adverse Bone Reactions | 6 months, 12 months, and 5 years
  Proportion of treated SIJs with adverse bone reactions at or near the SIJ.
Positive Bone Remodeling | 6 months, 12 months, and 5 years
  Proportion of treated SIJs with positive bone remodeling response.
SIJ Pain | Baseline, 3 mo, 6 mo, 12 mo, 24 mo, 60 months.
  Improvement from baseline in SIJ pain as measured by Visual Analog Scale
Disability | Baseline, 3 mo, 6 mo, 12 mo, 24 mo, 60 months.
  Improvement from baseline in disability as measured by Oswestry Disability Index.
QOL | Baseline, 3 mo, 6 mo, 12 mo, 24 mo, 60 months.
  Improvement from baseline in QOL as measured by EQ-5D
Physical Function | Baseline, 3 mo, 6 mo, 12 mo, 24 mo, 60 months.
  Improvement from baseline in physical function as measured by active straight leg raise, 5 times sit to stand, transitional timed up and go.
Opioid Use | Baseline, 3 mo, 6 mo, 12 mo, 24 mo, 60 months.
  Decrease from baseline in opioid use
Serious Adverse Event Rate | 3 mo, 6 mo, 12 mo, 24 mo, 60 months.
  Rate of serious adverse events related to the procedure or device.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Cher, MD, Study Director — SI-BONE, Inc.
Locations (11):
- United States (11):
  - Memorial Orthopaedic Surgical Group, Long Beach, California
  - University of Colorado Hospital, Aurora, Colorado
  - Clin Tech Center for Spine Health, Johnstown, Colorado
  - The B.A.C.K. Center, Melbourne, Florida
  - Orthopedic Center of Southern Illinois, Mount Vernon, Illinois
  - Bluegrass Orthopaedics, Lexington, Kentucky
  - LSU Health Sciences Center, Department of Neurosurgery, New Orleans, Louisiana
  - Columbia Orthopaedic Group, Columbia, Missouri
  - South Oregon Orthopedics, Medford, Oregon
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Aurora Research Institute, Green Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dat KO, Cher D, Polly DW. Effects of BMI on SI joint fusion outcomes: examining the evidence to improve insurance guidelines. Spine J. 2024 May;24(5):783-790. doi: 10.1016/j.spinee.2023.11.015. Epub 2023 Dec 9. PMID 38081463